CLINICAL TRIAL: NCT05108103
Title: How Far Should The Needle Be Withdrawn for Stellate Ganglion Block: Determination of Longus Colli Muscle Thickness by Ultrasonography
Brief Title: Determination of Longus Colli Muscle Thickness by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Halil Cetingok, Assistant Professor, Istanbul University
Other Study IDs: 2021/182
Record Dates: First submitted 2021-09-28; First posted 2021-11-04 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Pain Syndrome; Pain, Intractable; Complex Regional Pain Syndromes; Hyperhidrosis
Keywords: Stellate Ganglion; Longus Colli Muscle; Ultrasound
MeSH Terms: conditions — Somatoform Disorders; Pain, Intractable; Complex Regional Pain Syndromes; Hyperhidrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the longus colli muscle thickness by ultrasonography in order to guide stellate ganglion blocks

DETAILED DESCRIPTION:
Stellate ganglion block is an interventional pain management procedure that is often performed for diagnostic and therapeutic purposes. It has long been performed with the guidance of fluoroscopy, and despite the increasing use of ultrasonography in recent years, fluoroscopy is still the gold standard method.

In traditional fluoroscopic method, the needle is directed to the transverse process of the C6 vertebra, after touching the anterior tubercle (Chassaignac's tubercule) the needle is slightly withdrawn and following a negative aspiration, injection is performed.

The ideal placement of the needle should be anterolateral to the longus colli muscle and deep to the prevertebral fascia. Further placement may cause intramuscular spread and superficial placement may cause injection in the carotid sheath or vascular structures. These are the most important reasons for clinical ineffectiveness. How far should the needle be withdrawn? Data is inconsistent in the literature.

The primary aim of this study is to determine the distance from transverse process to longus colli muscles anterior border and from transverse process to carotid sheath's posterior border. Secondary aim is to investigate the relationship between longus colli muscle thickness and age, gender, height, weight, BMI and neck circumference.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 65 years,
* Giving informed consent for examination, ultrasonographic evaluation and study participation

Exclusion Criteria:

* Having a chronic neck pain for more than 6 months,
* Having any neurological or musculoskeletal conditions that may affect the anatomy of cervical region (cervical disc herniation, torticollis, severe scoliosis, vertebral malformation, spinal stenosis, myopathies, etc.)
* Having a history of surgery or radiation therapy in the cervical region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Distance between corpus and longus colli muscle's anterior border on C6 level (millimeters) | 0 minutes
  Distance between corpus and longus colli muscle's anterior border on C6 level will be evaluated with ultrasonography.

SECONDARY OUTCOMES:
Distance between corpus and longus colli muscle's anterior border on C7 level (millimeters) | 0 minutes
  Distance between corpus and longus colli muscle's anterior border on C7 level will be evaluated with ultrasonography.
Maximum anteroposterior width of longus colli muscle on C6 level (millimeters) | 0 minutes
  Maximum anteroposterior width of longus colli muscle on C6 level will be evaluated with ultrasonography.
Maximum anteroposterior width of longus colli muscle on C7 level (millimeters) | 0 minutes
  Maximum anteroposterior width of longus colli muscle on C6 level will be evaluated with ultrasonography.
Distance between esophagus and estimated needle plane (millimeters) | 0 minutes
  Distance between esophagus and estimated needle plane will be evaluated with ultrasonography.
Neck circumference (centimeters) | 0 minutes
  Neck circumference

CONTACTS AND LOCATIONS:
Overall Officials: Halil Çetingök, Ass. Prof., Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Pain Medicine
Locations (1):
- Halil Çetingök, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ates Y, Asik I, Ozgencil E, Acar HI, Yagmurlu B, Tekdemir I. Evaluation of the longus colli muscle in relation to stellate ganglion block. Reg Anesth Pain Med. 2009 May-Jun;34(3):219-23. doi: 10.1097/AAP.0b013e3181a32a02. PMID 19436184
- [Background] Narouze S. Ultrasound-guided stellate ganglion block: safety and efficacy. Curr Pain Headache Rep. 2014 Jun;18(6):424. doi: 10.1007/s11916-014-0424-5. PMID 24760493